CLINICAL TRIAL: NCT02755766
Title: Bracing Compliance and Personality Traits: A Compliance Assessment Program for Scoliosis and Clubfeet
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Henry J. Iwinski Jr., MD, Chief of Staff, Shriners Hospitals for Children
Other Study IDs: LEX-1501
Record Dates: First submitted 2016-03-28; First posted 2016-04-29 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Clubfeet; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Clubfeet: Babies, ages 0-1, with a diagnosis with clubfoot or clubfeet who are beginning treatment with foot abduction bracing following casting treatment.
- Adolescent Idiopathic Scoliosis: Patients, ages 10-14, with a diagnosis of AIS who are beginning treatment with TLSO (initial bracing).
- Guardians (CF babies): Clubfoot patients' guardians.

SUMMARY:
While studies have shown that better outcomes are associated with brace wear compliance in the scoliosis and clubfoot populations, compliance rates are still poor. Reasons identified by patients, parents and research for not complying with prescribed brace wear include the inconvenience or irritability of the child when in the brace in the case of clubfeet, and fear of looking different from peers, clothes not fitting properly, or discomfort in the case of scoliosis. While reasons for noncompliance are many and can be complex, there has been some research to indicate that personality traits may play a role in brace wear compliance.

The primary purpose of the proposed study is to determine if personality traits are related to compliance patterns for individuals undergoing brace treatment for AIS or Clubfeet.

DETAILED DESCRIPTION:
Bracing compliance, or the ability of patients to tolerate prescribed bracing regimens, has been shown to be related to the success of treatment. In pediatric orthopedics, bracing is used as one treatment option for a number of diagnoses and reasons. Two populations that are commonly prescribed bracing as part of the treatment paradigm are infants with clubfeet following Ponseti casting and adolescents with scoliosis.

For adolescents with idiopathic scoliosis, bracing is used to stop or slow progression of curves with the hope to delay or prevent the need for surgical intervention. Research has shown that bracing significantly decreased curve progression in patients with adolescent idiopathic scoliosis, and that the benefits of bracing increased with longer hours of brace wear.

Likewise, bracing is common practice for treating infants with clubfeet. All infants with clubfeet at SHC-Lexington are prescribed a bracing regimen following the completion of their Ponseti casting protocol. Previous research has shown that noncompliance with brace wear is strongly associated with recurrence of clubfeet in this population. Recurrence often leads to surgical intervention for these infants. Previous Kosair funded research conducted at SHC-Lexington investigated actual brace wear rates compared to the prescribed wear time in a sample of infants with clubfeet. In that study, brace wear rate significantly declined in the first three months of wear. That study did not look at factors related to the compliance with brace wear.

While studies have shown that better outcomes are associated with brace wear compliance in the scoliosis and clubfoot populations, compliance rates are still poor. Reasons identified by patients, parents and research for not complying with prescribed brace wear include the inconvenience or irritability of the child when in the brace in the case of clubfeet, and fear of looking different from peers, clothes not fitting properly, or discomfort in the case of scoliosis. While reasons for noncompliance are many and can be complex, there has been some research to indicate that personality traits may play a role in brace wear compliance. Work done by Rivett looked at personality traits of scoliotic girls who wore a Cheneau brace (a brace not commonly prescribed in North America and the United Kingdom) and found that those who were compliant with their bracing prescription tended to be more emotionally mature, stable and realistic than the noncompliant group. Although not well studied, personality traits of infants with clubfoot and their caregiver might similarly affect their compliance with brace wear.

Past work has shown that when braces are worn as prescribed, treatment outcomes are improved in those with scoliosis and clubfoot, yet bracing compliance is a consistent problem in both populations. With adolescent idiopathic scoliosis and clubfoot being the largest and third largest populations seen at SHC-Lexington, 3700 active patients and 2500 active patients, respectively, it is imperative that we address brace wear compliance in order to offer the best treatment outcome possible. At SHC-Lexington, during 2013 approximately 30 AIS patients and 50 infants with clubfoot were prescribed braces for the first time.

The primary purpose of the proposed study is to determine if personality traits are related to compliance patterns for individuals undergoing brace treatment for AIS or Clubfeet. This pilot project will examine different measures used to assess personality traits of adolescents with AIS, babies with clubfeet and their parent/guardian/caregiver. Using these identified measures, the association between traits and degree of compliance with the bracing prescriptions will be evaluated. If certain personality traits are identified as indicators for noncompliance, then additional support should be offered to those patients.

ELIGIBILITY:
Inclusion criteria for the clubfoot participants include:

* Less than a year of age
* Diagnosis of congenital clubfoot (unilateral or bilateral)
* Beginning treatment with foot abduction bracing following casting treatment

Exclusion criteria for the clubfoot participants include:

* Other diagnosis in addition to clubfoot
* Previous foot abduction bracing, and previous surgical correction (excluding tenotomy)

Exclusion criteria for the clubfoot guardians include:

* Under the age of 18 years
* Does not speak English

Inclusion for the AIS participants includes:

* Patients ages 10-14 years old
* Diagnosis of adolescent idiopathic scoliosis
* Beginning treatment with TLSO (initial bracing), and able to read
* Understand study questionnaires

Exclusion criteria for the AIS participants include:

* Other diagnosis in addition to AIS
* Previously prescribed brace for treatment

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 105 participants will be enrolled in the study. Of those 105, 35 will be clubfoot patients, 35 clubfoot patients' guardians, and 35 AIS patients.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2015-05-06 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Clubfoot brace compliance via iButton temperature monitor | 3 months
  Study Personnel will monitor brace wear using an iButton temperature monitor molded within the Dennis Browne brace. Orthotics personnel will place the sensor in the brace at the time of fabrication.
  Study Personnel will record if the participant was compliant with the 23 hours a day prescribed wear requirements and download the iButton data.
Scoliosis brace compliance via iButton temperature monitor | 6 months
  Study Personnel will monitor brace wear using an iButton temperature monitor molded within the TLSO. Orthotics personnel will place the sensor in the brace at the time of fabrication.
  Study Personnel will record if the participant was compliant with the 23 hours a day prescribed wear requirements and download the iButton data.

SECONDARY OUTCOMES:
Personality Assessment Guardian NEO-FFI-3 | 0 months
  The NEO Five Factor Inventory-3 (NEO-FFI-3) is a measure of the five domains of personality: neuroticism, extraversion, openness to experience, agreeableness, and conscientiousness. Guardians will complete this 60 item questionnaire at the initial visit.
Personality Assessment Baby IBQ-R Very Short | 3 months
  The Infant Behavior Questionnaire-Revised (IBQ-R) Very Short Form will be completed by the guardian to measure infant temperament. The form contains 36 items that measure 3 broad scales of temperament: surgency, negative affect, and effortful control.
Personality Assessment Adolescent FPPI-C | 0 months
  The Five Factor Personality Inventory (FPPI-C) is a measure of the five factors of personality: agreeableness, extraversion, openness to experience, conscientiousness, and emotional regulation. Participants will complete the 75 items on this assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Iwinski, MD, Principal Investigator — Shriners Hospital for Children
Locations (1):
- Shriners Hospital for Children, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No